CLINICAL TRIAL: NCT04634669
Title: An Open-Label Study to Assess the Long-term Safety and Efficacy of AXS-05 in Subjects With Treatment Resistant Depression
Brief Title: Open-Label Safety Study of AXS-05 in Subjects With TRD (EVOLVE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated once overall program objectives were met.
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXS-05-TRD-202
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
Keywords: AXS-05; Treatment Resistant Depression; TRD; NMDA receptor; Refractory depression; Resistant depression; Depression; Major depression; Dextromethorphan; Bupropion; MDD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AXS-05 (dextromethorphan-bupropion) (Experimental)
  Interventions: Drug: AXS-05 (dextromethorphan-bupropion)

INTERVENTIONS:
Drug: AXS-05 (dextromethorphan-bupropion) — - Titrated to AXS-05 (45 mg dextromethorphan HBr / 105 mg bupropion HCl) twice daily (up to 15 months)

SUMMARY:
This study is a multi-center, open-label trial to evaluate the long-term safety and efficacy of AXS-05 in subjects with major depressive disorder with prior treatment failures

DETAILED DESCRIPTION:
Eligible subjects must have either completed Study AXS-05-TRD-201 immediately prior to enrollment in this study or meet the DSM-5 criteria for major depressive disorder (MDD) without psychotic features.

ELIGIBILITY:
* Completed Study AXS-05-TRD-201 OR currently meets the DSM-5 criteria for MDD without psychotic features and with prior antidepressant treatment failure
* Agree to use adequate method of contraception for the duration of the study
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Chicago, Illinois
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, Staten Island, New York
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Raleigh, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, Friendswood, Texas
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Groups:
- AXS-05: AXS-05 tablet, taken twice daily (up to 15 months)
Period: Overall Study
Arm/Group | AXS-05
Started (Total number of subjects enrolled.) | 181
Completed (Number of subjects who Completed prior to study termination.) | 11
Not Completed | 170
Not completed — Study Terminated by Sponsor | 95
Not completed — Withdrawal by Subject | 20
Not completed — All Other Reasons | 55

BASELINE CHARACTERISTICS:
Arm/Group | AXS-05
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 144
  Black or African American | 29
  Asian | 3
  Other | 3
  Multiple | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent AEs (TEAEs) Following Dosing With AXS-05
Time Frame: Duration of participation was up to 15 months. TEAEs were defined as any AE with an onset date in the interval between the first study treatment dosing date and 7 days after the last study treatment dosing date.
Measure: Count of Participants; unit: Participants
Groups:
- AXS-05: AXS-05 tablet, taken twice daily for up to 15 months
Arm/Group | AXS-05
Number analyzed (Participants) | 181
Participants
  Subjects with any TEAEs | 112
  Subjects with suspected to be drug-related TEAEs | 65
  Subjects with serious TEAEs | 7
  Subjects with TEAEs that led to drug withdrawal | 16
  Subjects with TEAEs that led to withdrawal from study | 14
  Subjects with TEAEs that resulted in death | 0

ADVERSE EVENTS:
Time Frame: Duration of participation was up to 15 months. TEAEs were defined as any AE with an onset date in the interval between the first study treatment dosing date and 7 days after the last study treatment dosing date.
Arm/Group | AXS-05
All-Cause Mortality (participants affected / at risk) | 0/181
Serious Adverse Events (participants affected / at risk) | 7/181
Other Adverse Events (participants affected / at risk) | 38/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=181)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=181)
Covid-19 (Infections and infestations) | 15 (15)
Nausea (Gastrointestinal disorders) | 15 (15)
Headache (Nervous system disorders) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT04634669/Prot_001.pdf
  • Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT04634669/SAP_002.pdf